CLINICAL TRIAL: NCT05453292
Title: Feasibility, Safety, and Efficacy of EUS-guided Thermal Radiofrequency Ablation in the Treatment of Gastrointestinal Stromal Tumors
Brief Title: Endoscopic Ultrasound Radiofrequency Ablation for GISTs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IECED-05072022
Record Dates: First submitted 2022-07-05; First posted 2022-07-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: Gastrointestinal stromal tumor; Radiofrequency; Endosonography
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Intervention Model Description: A non-blinded, single center, non-randomized prospective feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS guided RFA (Experimental): This group is comprised by patients with diagnosis of resectable GISTs with/without liver metastasis. The patients included are naïve (without previous treatment) or patients with stable/progressive disease following systemic therapy with tyrosine kinase inhibitors.
  Interventions: Procedure: Endoscopic ultrasound guided radiofrequency ablation

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided radiofrequency ablation — Patients will be first assessed by DFI-EUS and CE-EUS. Then. EUS guided RFA will be performed using the 19G electrode ablation needle connected to the Starmed radiofrequency generator (Taewong Medical, Seoul, South Korea). After EUS identification of the GIST, a place without interposing vessels will be found by the endosonographer. Puncture of the tumor will be performed directly with the ablation probe inserted through the working channel of the echoendoscope. Time - seconds will depend by the tumor dimension, localization, distance from vital structures (e.g., aorta) and EUS appearance (e.g., hyperechoic). Power will be set at no more than 30W. If the tumor is in contact with vital structures a 10mm safe margin will be kept from these to avoid thermal injury. Multiple applications can be performed in the same or separate session depending on the residual tumor tissue evaluated with DFI-EUSor CE-EUS immediately after procedure.

SUMMARY:
Nowadays, for the selection of the treatment for gastrointestinal stromal tumors (GISTs), tumor size, prognosis, resectability and stage should be considered. Due to mutations in KIT and platelet-derived growth factor alpha (PDGFRA) in 90% of patients with this mesenchymal tumor, many tyrosine kinase inhibitors are used. On the other hand, a resectable tumor is approached by surgery, endoscopic and ablation therapy.

Radiofrequency ablation (RFA) approach has been studied in hepatic GISTs, and hepatic metastases, but its evaluation in esophageal, gastric, and intestinal GISTs is scarce. This study aims to determine the feasibility, safety and efficacy of endoscopic ultrasound (EUS) guided RFA using the 19 G RFA probe developed by Taewong Medical for the treatment of GISTs.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GISTs) are the most common malignant mesenchymal tumors of the gastrointestinal tract. GISTs usually appear like subepithelial lesions covered by normal mucosa, arising from the second of fourth layer of the gastrointestinal tract wall. They are variable in size and mostly asymptomatic, but they can present different clinical behavior as bleeding, pain, or obstruction. The tumor size, location and mitotic rate are important prognostic factors. For resectable tumors >2 cm, surgery is the treatment of choice; the management of tumors <2 cm remains debatable because they present unclear clinical significance and low risk of malignancy. Endoscopic treatment, when complete resection it's possible, could be an option to full thickness laparoscopic resection. Moreover, around 90% of GISTs harbour driver mutation in KIT and platelet-derived growth factor alpha (PDGFRA), making the treatment with tyrosine kinase inhibitors (i.e., imatinib, sunitinib and regorafenib) a suitable option for locally advanced and metastatic disease. Nevertheless, the role of local treatment in advanced and metastatic disease is limited, with few retrospective studies suggesting tumor ablation as a therapeutic approach.

According to literature, thermal ablation has been successfully used for local treatment of hepatic metastases from GISTs (as a curative treatment). However, its feasibility and technical success as a local treatment in esophageal, gastric or intestinal GISTs has not been evaluated.

The investigators aimed to determine the feasibility and efficacy of the RFA electrode developed by Taewong Medical for the treatment of resectable GISTs (esophageal, gastric and intestinal lesions) as well as its limited liver metastases in naïve patients or patients with stable disease following systemic therapy with tyrosine kinase inhibitors. The challenge is whether to introduce local ablative therapy as curative or as part of multimodal treatment in patients with GISTs to obtain a curable disease and an increase in overall survival for metastatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years of age)
* Confirmed resectable GISTs lesions in esophagus, stomach, and intestine (between 2<5 cm or 5-10cm and <5mitotes/HPF)
* Non-amenable to surgery
* written informed consent
* No evidence of metastatic disease on imaging of the chest abdomen and pelvis contrast enhanced computed tomography (CE-CT) or limited liver metastatic disease (maximum 5 lesions <= 3 cm)
* Adequate renal, hepatic, and hematological function

Exclusion Criteria:

* Pregnancy
* Rectal GISTs
* Altered renal, hepatic, or hematological function
* Inability to provide informed consent
* Patients with cardiac pacemakers or other implanted electronic devices and/or electrodes
* Patients that have right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension, and in patients with adult respiratory distress syndrome or any condition that contraindicates the procedure
* Inability to tolerate general anesthesia.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 6 months
  Incidence of adverse events of EUS guided RFA for GISTs' lesions and metastasis. Data will be summarized as frequencies and relative frequencies.
Technical success of RFA of GISTs lesions and metastasis | up to 2 hours
  The technical success will be assessed by completion of ablation on EUS by the time of the procedure, indicated by replacement of the lesion by structural/appearance changes on DFI and CE-EUS Data will be summarized as frequencies.
Disease-free survival | up to 6 months
  Will be assessed by measuring the proportion of patients demonstrating absence of residual tumor on follow-up. CT- scan and DFI at one, three and six months will be performed to evaluate tumor response to the treatment.
  Will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% confidence intervals.

SECONDARY OUTCOMES:
Re-treatment rate | 1-month
  Proportion of patients needing re-treatment for residual tumor in a one-month period after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Farag S, Smith MJ, Fotiadis N, Constantinidou A, Jones RL. Revolutions in treatment options in gastrointestinal stromal tumours (GISTs): the latest updates. Curr Treat Options Oncol. 2020 May 27;21(7):55. doi: 10.1007/s11864-020-00754-8. PMID 32462367
- [Background] Casali PG, Blay JY, Abecassis N, Bajpai J, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brodowicz T, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dufresne A, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Frezza AM, Gasperoni S, Gelderblom H, Gouin F, Grignani G, Haas R, Hassan AB, Hindi N, Hohenberger P, Joensuu H, Jones RL, Jungels C, Jutte P, Kasper B, Kawai A, Kopeckova K, Krakorova DA, Le Cesne A, Le Grange F, Legius E, Leithner A, Lopez-Pousa A, Martin-Broto J, Merimsky O, Messiou C, Miah AB, Mir O, Montemurro M, Morosi C, Palmerini E, Pantaleo MA, Piana R, Piperno-Neumann S, Reichardt P, Rutkowski P, Safwat AA, Sangalli C, Sbaraglia M, Scheipl S, Schoffski P, Sleijfer S, Strauss D, Strauss SJ, Hall KS, Trama A, Unk M, van de Sande MAJ, van der Graaf WTA, van Houdt WJ, Frebourg T, Gronchi A, Stacchiotti S; ESMO Guidelines Committee, EURACAN and GENTURIS. Electronic address: clinicalguidelines@esmo.org. Gastrointestinal stromal tumours: ESMO-EURACAN-GENTURIS Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2022 Jan;33(1):20-33. doi: 10.1016/j.annonc.2021.09.005. Epub 2021 Sep 21. No abstract available. PMID 34560242
- [Background] Yamashita Y, Yoshikawa T, Kawaji Y, Tamura T, Hatamaru K, Itonaga M, Ida Y, Maekita T, Iguchi M, Murata SI, Kitano M. Novel endoscopic ultrasonography imaging technique for visualizing microcirculation without contrast enhancement in subepithelial lesions: Prospective study. Dig Endosc. 2021 Sep;33(6):955-961. doi: 10.1111/den.13889. Epub 2020 Dec 23. PMID 33145842
- [Background] Yamashita Y, Yoshikawa T, Yamazaki H, Kawaji Y, Tamura T, Hatamaru K, Itonaga M, Ashida R, Ida Y, Maekita T, Iguchi M, Kitano M. A Novel Endoscopic Ultrasonography Imaging Technique for Depicting Microcirculation in Pancreatobiliary Lesions without the Need for Contrast-Enhancement: A Prospective Exploratory Study. Diagnostics (Basel). 2021 Oct 30;11(11):2018. doi: 10.3390/diagnostics11112018. PMID 34829364
- [Background] Granata V, Grassi R, Fusco R, Setola SV, Palaia R, Belli A, Miele V, Brunese L, Grassi R, Petrillo A, Izzo F. Assessment of Ablation Therapy in Pancreatic Cancer: The Radiologist's Challenge. Front Oncol. 2020 Nov 27;10:560952. doi: 10.3389/fonc.2020.560952. eCollection 2020. PMID 33330028
- [Background] Robles-Medranda C, Arevalo-Mora M, Oleas R, Alcivar-Vasquez J, Del Valle R. Novel EUS-guided microwave ablation of an unresectable pancreatic neuroendocrine tumor. VideoGIE. 2022 Jan 19;7(2):74-76. doi: 10.1016/j.vgie.2021.10.009. eCollection 2022 Feb. PMID 35146230
- [Background] Yamanaka T, Takaki H, Nakatsuka A, Uraki J, Fujimori M, Hasegawa T, Sakuma H, Yamakado K. Radiofrequency ablation for liver metastasis from gastrointestinal stromal tumor. J Vasc Interv Radiol. 2013 Mar;24(3):341-6. doi: 10.1016/j.jvir.2012.11.021. Epub 2013 Jan 24. PMID 23352855